CLINICAL TRIAL: NCT05057793
Title: A Prospective, Multicentre, Randomised, Assessor Blinded Study Comparing the Efficacy, Including Participant Reported Outcomes, of Daily Geko™ Therapy in Conjunction With Standard Care to Standard Care Alone, in Patients With Venous Leg Ulcers
Brief Title: Efficacy Study for Geko Device in VLU Patients (Canada)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with recruitment
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSK-VLU-006
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Venous Leg Ulcer; Leg Ulcer; Venous Ulcer
Keywords: geko; compression bandaging; wound; ulcer
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer; Wounds and Injuries; Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Multilayer, multicomponent compression intended for the treatment of VLU
- Standard of care + geko 12h (Active Comparator): Multilayer multicomponent compression intended for the treatment of VLU in conjuction with geko™ therapy 12 hours daily
  Interventions: Device: geko

INTERVENTIONS:
Device: geko — The geko device will be self-administered and deliver 12 hours of therapy daily.
  Other Names: NMES; geko device; geko 12h
  Arms: Standard of care + geko 12h

SUMMARY:
The objective of this study is to compare the efficacy of a daily geko™ wound therapy (duration of 12 hours), in conjunction with standard of care (SC), to SC alone, in participants with venous leg ulcers.The participants will go through a four-week run-in phase, followed by a four-week treatment phase and a three-month long term follow-up.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy of geko™ therapy for 12 hours daily in conjunction with Standard Care (SC), consisting of multilayer, multicomponent compression therapy intended for the treatment of VLUs, compared to SC alone in participants with VLUs.

The study will be a multicentre study with study centres in Ontario Canada.

The study will have three phases:

1. A four-week Run-In Phase (day 0-28)
2. A four-week Treatment Phase (day 28-56)
3. A long term Follow-Up Phase (day 84, 112 & 140 after EOT)

During the Run-In Phase all participants will receive SC only and will be evaluated on a weekly basis (day 0, 7, 14 & 21). On day 28, once the Investigator has confirmed the participant's continued eligibility, randomization and assignment to study treatment will take place. During the long term follow-up phase, participants continue with their assigned study treatment and will be seen and evaluated on day 84, 112 and 140

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years, able to provide written informed consent and comply with all study procedures and visit schedule
2. Intact healthy skin at the site of geko™ device application.
3. Have a (chronic) venous leg ulcer determined to be due to underlying venous disease following evaluation in a multi-professional setting or by a vascular surgeon, specialist physician or nurse wound specialist in accordance with Wounds Canada (2018), Health Quality Ontario Standards
4. A VLU of approximately ≥ 5cm2 and ≤ 40cm2 at study enrolment i.e. Run in Phase Visit 1. If more than one ulcer is present, the largest ulcer within the given size range will be designated the study ulcer and the only one included in the study. If other ulcerations are present on the same leg, they must be more than 2 cm apart if they are two separate wounds.
5. Study ulcer (current episode of ulceration in case of ulcer recurrence) has been present for at least 6 weeks but no more than 5 years prior to study entry.
6. Ankle-Brachial Pressure Index (ABPI) of 0.8 -1.2 ± 0.05 inclusive (or equivalent measure) measured at study entry or within 12 weeks of study entry.
7. No active local index wound infection for a minimum of 48 hours prior to study entry (RV1)
8. No systemic antimicrobial treatment for a minimum of seven days prior to study entry (RV1) prescribed for index wound infection
9. Must understand and is willing and able to participate in the study and to comply with all study procedures and study visit schedule

Exclusion Criteria:

1. Known allergy or intolerance to any of the protocol-stipulated treatments
2. History of significant haematological disorders (e.g. Sickle Cell disease)
3. History of Deep Vein Thrombosis (DVT) within six months preceding study entry
4. History of Pyoderma Gangrenosum or other inflammatory ulceration
5. BMI ≥ 40
6. Pregnancy or risk of pregnancy
7. Use of investigational drug or device within four weeks prior to study entry that may interfere with the study
8. Use of any neuro-modulation device
9. Surgery during three months prior to study entry (such as abdominal, gynaecological, hip or knee replacement)
10. Trauma to the lower limbs that would prevent geko™ from stimulating the common peroneal nerve.
11. Implanted with a pacemaker or implantable cardioverter defibrillator (ICD).
12. Any medication deemed by the Investigator to potentially interfere with the study treatment (e.g. higher dose systemic steroids).
13. Participation in any other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Change in linear healing rate in the treatment phase compared to the run-in phase | 8 weeks
  The pair-wise comparison of linear healing rate (wound margin advance, WMA) during Treatment Phase compared with WMA from the Run-in Phase both the treatment arm (SC plus 12 hours daily treatment with the geko™ W device or variant) and control arm (SC only).

SECONDARY OUTCOMES:
Weekly change in linear healing rate | 8 weeks
  Weekly wound margin advance of the study ulcer measured by an independent blinded wound expert using digital images taken at each weekly visit until end of treatment.
Change in pain score using the VAS (Visual Analogue Scale) | 8 weeks
  Patient will indicate their pain score at each weekly visit using a visual analogue scale (VAS), with 0 being no pain at all and 100 being worst pain imaginable (measured in mm)
Change in quality of life using the EQ-5D-5L (health-related quality of life measure) questionnaire | 8 weeks
  EQ-5D-5L a descriptive system for health-related quality of life (HRQoL) states in adults, consisting of five dimensions (mobility, self-care, usual activities, pain & discomfort, anxiety & depression). Participant will complete questionnaire at the beginning of the run in phase, at randomization and at the end of treatment. Each level is scored ona 5 level severity ranking, with 1 being no problems, to 5 being extreme problems.
Change in quality of life using the CWIS (Cardiff Wound Impact Schedule) | 8 weeks
  Cardiff Wound Impact Schedule (CWIS) is used to measure the impact of chronic wounds (leg ulcers and diabetic foot ulcers) on HRQoL and identify areas of participant concern. The questionnaire will be completed by the participant at the beginning of the run in phase, at randomization and at the end of treatment. The overall score will be between 0 and 100, with a higher score indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Garry Sibbald, Principal Investigator — University of Toronto
Locations (3):
- Canada (3):
  - The Mayer Institute, Hamilton
  - Vascular Health Bronte, Oakville
  - Care Partners (Waterloo), Waterloo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Device official website — https://www.gekodevices.com/